CLINICAL TRIAL: NCT02426931
Title: Tip-flexible Semi-rigid Ureterorenoscope Versus Flexible Ureteroscopy for the Treatment of Renal Calculi < 3 cm - Efficacity Prospective Randomized Multicentre Trial
Brief Title: Tip-flexible Semi-rigid Ureterorenoscope Versus Flexible Ureteroscopy in Renal Calculi
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ling Li, MD (Other)
Collaborators: Changhai Hospital (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); Xiangya Hospital of Central South University (Other); Ningbo No. 1 Hospital (Other); West China Hospital (Other); Beijing Tsinghua Changgeng Hospital (Other); Yantai Yuhuangding Hospital (Other)
Responsible Party: Sponsor-Investigator, Ling Li, MD, Chief of Department of Urology, Changhai Hospital
Organization: Changhai Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01
Record Dates: First submitted 2015-02-12; First posted 2015-04-27 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2015-04

CONDITIONS: Renal Calculi
Keywords: retrograde intrarenal surgery; flexible ureteroscopy; renal calculi
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tf-URS (Experimental): Participants in tf-URS group undergo ureteroscopy using the tip-flexible ureterorenoscope.
  Interventions: Device: the tip-flexible ureterorenoscope
- f-URS (Active Comparator): Participants in f-URS group undergo ureteroscopy using the classic flexible ureteroscope.
  Interventions: Device: the classic flexible ureteroscope

INTERVENTIONS:
Device: the tip-flexible ureterorenoscope — Ureteroscopy will be conducted using the tip-flexible semi-rigid ureterorenoscope to treat renal calculi. Holmium laser and basket can be used to perform the technique.
  Arms: tf-URS
Device: the classic flexible ureteroscope — Ureteroscopy will be conducted using the classic flexible ureteroscope (Flex x2 STORZ, Germany) to treat renal calculi. Holmium laser and basket can be used to perform the technique.
  Arms: f-URS

SUMMARY:
This study evaluates the safety and efficacy of the novel tip-flexible semi-rigid ureterorenoscope for the treatment of renal calculi using a prospective, randomized multicentre trial design. Half of participants will receive retrograde intrarenal surgery using the tip-flexible semi-rigid ureterorenoscope, while the other half participants will receive retrograde intrarenal surgery using the classic flexible ureteroscope.

DETAILED DESCRIPTION:
Retrograde intrarenal surgery using flexible ureteroscope has become the first-line treatment for renal calculi < 3.0 cm and is recommended by the European Association of Urology due to its minimally-invasive nature and satisfactory result.

However, some limitations still remain. Poor maneuverability, extra costs for the ureteral access sheath, and high device vulnerability still preclude flexible ureteroscopy from wider distribution.

Recently, the investigators present a novel ureterorenoscope, which is composed of a retractable rigid sheath and a semi-rigid ureteroscope with a flexible part on the tip. When the flexible tip of the inner shaft maintains within the sheath, working in the "rigid mode", the tip-flexible semi-rigid ureterorenoscope is capable of passing either the orifice or the physiological tortuosity of the ureter with ease. When the inner shaft is extended beyond the sheath, the endoscope is switched to the "flexible mode", capable of performing an intrarenal approach.

This endoscope integrates the classic semi-rigid and flexible ureteroscope both structurally and functionally, and has been approved for clinical application by the China Food and Drug Administration. In this study, transverse comparison is designed to evaluate the safety and efficacy of the tip-flexible semi-rigid ureterorenoscope for the treatment of renal calculi.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent and indicated a willingness to comply with study treatments
* Subject has a diagnosis of renal stones according to computer tomography (CT) and intravenous pyelogram (IVP) results
* Subject is a surgical candidate for the ureteroscopic approach
* Subject is 18-80 yrs of age
* Subject has a single stone < 3 cm in size (IVP), or multiple stones < 3 cm in cumulative size (IVP)
* Subject has a serum creatinine level within the normal range for the study center

Exclusion Criteria:

* Subject needs bilateral procedures within one-stage ureteroscopy
* Subject has an active urinary tract infection (e.g., cystitis, prostatitis, urethritis, etc.)
* Subject has been diagnosed with a urethral stricture or bladder neck contracture
* Subject has been diagnosed with a urinary tract infection related to stone obstruction within two weeks
* Subject has severe hematuria that might blur the vision of the endoscopy
* Subject has a disorder of the coagulation cascade system that would put the subject at risk for intraoperative or postoperative bleeding
* Subject is unable to discontinue anticoagulant and antiplatelet therapy preoperatively (3-5 d)
* Subject has other diseases and could not tolerate the endoscopic surgery
* Subject has any kind of anatomic abnormality of the urinary system that might have an influence on the surgery
* Subject has ipsilateral pre-stenting or previous ureteroscopy within six months
* Subject has been diagnosed with hydronephrosis larger than 3 cm according to the B-scan ultrasonography examination

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Stone clearance | 12 weeks post-operatively
  Number of participants undergo tf-URS or f-URS surgeries without residual calculus/Total number of participants in each group *100%

SECONDARY OUTCOMES:
Stone clearance | One day post-operatively
  Number of participants undergo tf-URS or f-URS surgeries without residual calculus/Total number of participants in each group *100%
Complication rates | Within 12 weeks after surgery
  Number of participants undergo tf-URS or f-URS surgeries suffer complications associated with the surgery (i.e. painess(NRS≥4), hematuria, T≥38℃, serum WBC≥12×〖10〗^9/L ,serum WBC<4×〖10〗^9/L, perforation, etc.)/Total number of participants in each group *100%
Endoscope deflection loss rates | intraoperative
  Number of the broken novel ureterorenoscope or the broken classic flexible ureterosocpe with deflection loss>10%/Total number of ureterorenoscope or ureterosocpe used *100%
Endoscope Leakage rates | intraoperative
  Number of the broken novel ureterorenoscope or the broken classic flexible ureterosocpe with leakage of the working channel or the outer shaft/times of the ureterorenoscope or ureterosocpe used *100%
Endoscope black dots rates | intraoperative
  Number of the broken novel ureterorenoscope or the broken classic flexible ureterosocpe with black dots on endoscopic images/times of ureterorenoscope or ureterosocpe used *100%

CONTACTS AND LOCATIONS:
Overall Officials: Yinghao Sun, MD, Study Chair — Changhai Hospital; Guohua Zeng, MD, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University; Hequn Chen, MD, Principal Investigator — Xiangya Hospital of Central South University; Yue Cheng, MD, Principal Investigator — Ningbo No. 1 Hospital; Kunjie Wang, MD, Principal Investigator — West China Hospital; Jianxing Li, MD, Principal Investigator — Beijing Tsinghua Changgeng Hospital; Lei Shi, MD, Principal Investigator — Yantai Yuhuangding Hospital; Xiaofeng Gao, MD, Principal Investigator — Changhai Hospital

REFERENCES:
- [Background] Aboumarzouk OM, Monga M, Kata SG, Traxer O, Somani BK. Flexible ureteroscopy and laser lithotripsy for stones >2 cm: a systematic review and meta-analysis. J Endourol. 2012 Oct;26(10):1257-63. doi: 10.1089/end.2012.0217. Epub 2012 Jul 30. PMID 22642568
- [Background] de la Rosette J, Denstedt J, Geavlete P, Keeley F, Matsuda T, Pearle M, Preminger G, Traxer O; CROES URS Study Group. The clinical research office of the endourological society ureteroscopy global study: indications, complications, and outcomes in 11,885 patients. J Endourol. 2014 Feb;28(2):131-9. doi: 10.1089/end.2013.0436. Epub 2013 Dec 17. PMID 24147820
- [Background] Geavlete P, Multescu R, Geavlete B. Pushing the boundaries of ureteroscopy: current status and future perspectives. Nat Rev Urol. 2014 Jul;11(7):373-82. doi: 10.1038/nrurol.2014.118. Epub 2014 Jun 3. PMID 24890883
- [Background] Yoon PD, Chalasani V, Woo HH. Use of Clavien-Dindo classification in reporting and grading complications after urological surgical procedures: analysis of 2010 to 2012. J Urol. 2013 Oct;190(4):1271-4. doi: 10.1016/j.juro.2013.04.025. Epub 2013 Apr 11. PMID 23583859
- [Background] Yinghao S, Yang B, Gao X. The management of renal caliceal calculi with a newly designed ureteroscope: a rigid ureteroscope with a deflectable tip. J Endourol. 2010 Jan;24(1):23-6. doi: 10.1089/end.2009.0030. PMID 20059383
- [Background] Rebuck DA, Macejko A, Bhalani V, Ramos P, Nadler RB. The natural history of renal stone fragments following ureteroscopy. Urology. 2011 Mar;77(3):564-8. doi: 10.1016/j.urology.2010.06.056. Epub 2010 Dec 15. PMID 21109293
- [Background] Traxer O, Thomas A. Prospective evaluation and classification of ureteral wall injuries resulting from insertion of a ureteral access sheath during retrograde intrarenal surgery. J Urol. 2013 Feb;189(2):580-4. doi: 10.1016/j.juro.2012.08.197. Epub 2012 Oct 8. PMID 22982421
- [Background] Atis G, Arikan O, Gurbuz C, Yildirim A, Erol B, Pelit S, Ulus I, Caskurlu T. Comparison of different ureteroscope sizes in treating ureteral calculi in adult patients. Urology. 2013 Dec;82(6):1231-5. doi: 10.1016/j.urology.2013.07.021. Epub 2013 Sep 12. PMID 24035032
- [Background] Perez Castro E, Osther PJ, Jinga V, Razvi H, Stravodimos KG, Parikh K, Kural AR, de la Rosette JJ; CROES Ureteroscopy Global Study Group. Differences in ureteroscopic stone treatment and outcomes for distal, mid-, proximal, or multiple ureteral locations: the Clinical Research Office of the Endourological Society ureteroscopy global study. Eur Urol. 2014 Jul;66(1):102-9. doi: 10.1016/j.eururo.2014.01.011. Epub 2014 Jan 23. PMID 24507782
- [Background] Karadag MA, Demir A, Cecen K, Bagcioglu M, Kocaaslan R, Altunrende F. Flexible ureterorenoscopy versus semirigid ureteroscopy for the treatment of proximal ureteral stones: a retrospective comparative analysis of 124 patients. Urol J. 2014 Nov 1;11(5):1867-72. PMID 25361706
- [Background] Wendt-Nordahl G, Mut T, Krombach P, Michel MS, Knoll T. Do new generation flexible ureterorenoscopes offer a higher treatment success than their predecessors? Urol Res. 2011 Jun;39(3):185-8. doi: 10.1007/s00240-010-0331-0. Epub 2010 Nov 5. PMID 21052986
- [Background] Wendt-Nordahl G, Trojan L, Alken P, Michel MS, Knoll T. Ureteroscopy for stone treatment using new 270 degrees semiflexible endoscope: in vitro, ex vivo, and clinical application. J Endourol. 2007 Dec;21(12):1439-44. doi: 10.1089/end.2006.0291. PMID 18186680
- [Background] Geavlete P, Multescu R, Geavlete B. Retrograde flexible ureteroscopic approach of upper urinary tract pathology: What is the status in 2014? Int J Urol. 2014 Nov;21(11):1076-84. doi: 10.1111/iju.12582. Epub 2014 Aug 1. PMID 25081354
- [Background] Bedke J, Leichtle U, Lorenz A, Nagele U, Stenzl A, Kruck S. 1.2 French stone retrieval baskets further enhance irrigation flow in flexible ureterorenoscopy. Urolithiasis. 2013 Apr;41(2):153-7. doi: 10.1007/s00240-012-0540-9. Epub 2013 Jan 5. PMID 23503877
- [Background] Somani BK, Al-Qahtani SM, de Medina SD, Traxer O. Outcomes of flexible ureterorenoscopy and laser fragmentation for renal stones: comparison between digital and conventional ureteroscope. Urology. 2013 Nov;82(5):1017-9. doi: 10.1016/j.urology.2013.07.017. Epub 2013 Aug 31. PMID 24001703
- [Background] Ozsoy M, Acar O, Sarica K, Saratlija-Novakovic Z, Fajkovic H, Librenjak D, Esen T, Scheffbuch N, Seitz C. Impact of gender on success and complication rates after ureteroscopy. World J Urol. 2015 Sep;33(9):1297-302. doi: 10.1007/s00345-014-1435-x. Epub 2014 Nov 12. PMID 25385490